CLINICAL TRIAL: NCT03777566
Title: Uterine Cavity Volume Measuring With Sonohysterography: A New Objective Method
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mohamed I Amer, Professor, Ain Shams University
Other Study IDs: mohamed amer
Record Dates: First submitted 2018-12-14; First posted 2018-12-17 (Actual); Last update posted 2019-12-23 (Actual); Status verified 2019-12

CONDITIONS: Cavity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group A: 35 patients with an indication for hysterectomy without gross uterine pathology
  Interventions: Diagnostic Test: sonohysterography
- group B: 150 infertile patients in the childbearing age without gross uterine pathology
  Interventions: Diagnostic Test: sonohysterography

INTERVENTIONS:
Diagnostic Test: sonohysterography — sonohysterography with measuring the uterine cavity volume

SUMMARY:
Measuring of uterine cavity volume using sonohysterography will be done in two groups of patients, Group A included 35 patients for home hysterectomy were indicated and group B includes 150 infertile patients in the childbearing age.

DETAILED DESCRIPTION:
Uterine cavity volume will be measured in group A before and after hysterectomy, and in the group, B will be measured using sonohysterography only using a mathematical method of the sum of a volume of a cone and part of a sphere.

ELIGIBILITY:
Inclusion Criteria:

1. Patients without any gross pathology within the uterus.
2. Patients admitted for hysterectomy.
3. Patients agreed with written consent to participate in the study.

Exclusion Criteria:

1. Virgins.
2. Pregnancy.
3. Systemic blood disease.
4. Any clinical evidence of cervical, uterine or tubal infection.
5. Refusal to undergo saline infusion sonography.
6. Any gross uterine pathology diagnosed clinically or with sonography.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Women undergo sonohysterography for gynecologic indication without gross uterine pathology.
Sampling Method: Non-Probability Sample
Enrollment: 185 (Estimated)
Dates: Start 2019-02-10 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
calculation of uterine cavity volume with an objective method | one day
  measuring uterine cavity volume objectively

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed I Amer, MD, Principal Investigator — Ain Shams University
Locations (1):
- AIn Shams University Maternity Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No